CLINICAL TRIAL: NCT04706546
Title: Hemodynamic Effects of Acute Normobaric Hypoxia During Exercise in Patients With Pulmonary Hypertension: Single-center Randomized Controlled Trial
Brief Title: Hemodynamic Effects During Exercise in Patients With Pulmonary Hypertension Receiving Sildenafil
Acronym: HEXASN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 2020-02163_A2
Record Dates: First submitted 2020-12-20; First posted 2021-01-13 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2022-05

CONDITIONS: Hypertension, Pulmonary
Keywords: hypoxia; exercise; hemodynamics; Vasodilative drug
MeSH Terms: conditions — Hypertension, Pulmonary; Hypoxia; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemodynamic effect of exercise under Sildenafil (Experimental): Inhalation of room air through an altitude simulator ("Altitrainer"), for approx. 1/2 hour given by a facemask, first at rest and then during exercise under SIldenafil.
  Interventions: Other: Hemodynamic effect of exercise under Sildenafil
- Hemodynamic effect of exercise (Other): Inhalation of room air through an altitude simulator ("Altitrainer"), for approx. 1/2 hour given by a facemask, first at rest and then during exercise.
  Interventions: Other: Hemodynamic effect of exercise

INTERVENTIONS:
Other: Hemodynamic effect of exercise under Sildenafil — Inhalation of room air through an altitude simulator ("Altitrainer"), for approx. 1/2 hour given by a facemask, first at rest and then during exercise under SIldenafil.
  Arms: Hemodynamic effect of exercise under Sildenafil
Other: Hemodynamic effect of exercise — Inhalation of room air through an altitude simulator ("Altitrainer"), for approx. 1/2 hour given by a facemask, first at rest and then during exercise.
  Arms: Hemodynamic effect of exercise

SUMMARY:
To study hemodynamic effects of Sildenafil during exercise in patients with pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent as documented by signature (Appendix Informed Consent Form)
* PH class I (PAH) or IV (CTEPH) diagnosed according to guidelines: mean pulmonary artery pressure >20 mmHg, pulmonary vascular resistance ≥3 wood units, pulmonary arterial wedge pressure ≤15 mmHg during baseline measures at the diagnostic right-heart catheterization

Exclusion Criteria:

* resting partial pressure of oxygen <8 kilopascal at Zürich altitude on ambient air
* exposure to an altitude >1000 m for ≥3 nights during the last 2 weeks before the study
* inability to follow the procedures of the study
* patients who take nitrates
* other clinically significant concomitant end-stage disease (e.g., renal failure, hepatic dysfunction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
mean pulmonary artery pressure (mPAP) / cardiac output (CO) | 4 hours
  Difference in mPAP/CO during exercise between tests under normoxia with/without Sildenafil

SECONDARY OUTCOMES:
Differences in pulmonary arterial pressure | 4 hours
  Differences in pulmonary arterial pressure at rest and during exercise under normoxia with/without Sildenafil
Differences in cardiac output | 4 hours
  Differences in cardiac output at rest and during exercise under normoxia with/without Sildenafil
Differences in pulmonary vascular resistance | 4 hours
  Differences in pulmonary vascular resistance at rest and during exercise under normoxia with/without Sildenafil
Differences in pulmonary artery wedge pressure | 4 hours
  Differences in pulmonary artery wedge pressure at rest and during exercise under normoxia with/without Sildenafil
Differences in right atrial pressure | 4 hours
  Differences in right atrial pressure at rest and during exercise under normoxia with/without Sildenafil
Differences in mixed venous oxygen saturation | 4 hours
  Differences in mixed venous oxygen saturation at rest and during exercise under normoxia with/without Sildenafil
Differences in heart rate | 4 hours
  Differences in heart rate at rest and during exercise, under normoxia with/without Sildenafil
Differences in blood pressure (systolic and diastolic) | 4 hours
  Differences in blood pressure (systolic and diastolic) at rest and during exercise, under normoxia with/without Sildenafil
Differences in oxygen saturation | 4 hours
  Differences in oxygen saturation at rest and during exercise, under normoxia with/without Sildenafil
Differences in arterial blood gases | 4 hours
  Differences in arterial blood gases at rest and during exercise under normoxia with/without Sildenafil
Differences in mixed venous blood gases | 4 hours
  Differences in mixed venous blood gases at rest and during exercise under normoxia with/without Sildenafil
Differences in cerebral tissue oxygenation | 4 hours
  Differences in cerebral tissue oxygenation at rest and during exercise, under normoxia with/without Sildenafil
Differences in muscle tissue oxygenation | 4 hours
  Differences in muscle tissue oxygenation at rest and during exercise, under normoxia with/without Sildenafil
Differences in symptoms (Borg dyspnoea) | 4 hours
  Differences in symptoms (Borg dyspnoea, Borg CR10, scale 0-10) at rest and during exercise under normoxia with/without Sildenafil
Differences in symptoms (leg effort) | 4 hours
  Differences in symptoms (leg effort, scale 0-10, 10 is maximal exhaustion) at rest and during exercise under normoxia with/without Sildenafil

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Ulrich, Prof. Dr., Principal Investigator — UniversityHospital Zurich, Department of Pulmonology
Locations (2):
- Switzerland (2):
  - University Hospital of Zurich, Zurich, Canton of Zurich
  - UniversityHospital Zurich, Department of Pulmonology, Zurich

IPD SHARING:
Plan to Share IPD: Yes
We will share individual participant data after publication of the manuscript. The decision about the platform is ongoing.
Time Frame: After publication of the manuscript.